CLINICAL TRIAL: NCT04302285
Title: Impact of Single Exercise Session Conducted Prior to Phenylketonuria (PKU) Type Meal on Appetite Hormones, Metabolic Rate, Fat Oxidation and Energy Intake
Brief Title: Impact of Single Exercise Session Conducted Prior to PKU Type Meal on Appetite Hormones and Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Dalia Malkova, Dr, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 200170151
Record Dates: First submitted 2020-02-04; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise trial (Experimental): In this trial, participants were asked to exercise for one hour under controlled laboratory conditions. Participants were exercising on the treadmill at speed and grade corresponding to 60% of their V̇O2max. Participants were wearing a HR monitor and a face mask while exercising, connected to indirect calorimetry equipment. Appetite questionnaires were obtained, and blood samples were collected at 30, 60, 90 and 120 pre-meal, 150, 180, 210, 240 and 300 min post-meal. Metabolic rate was measured every 30 min after each blood sample. Participants were presented to a standard isocaloric PKU type meal at 120 min. After the completion of the last measurement, the participants were presented with an ad libitum buffet test meal.
  Interventions: Other: PKU type meal and Exercise
- Control trial (Experimental): In this trial, participants were asked to rest for one hour. Appetite questionnaires were obtained, and blood samples were collected at 30, 60, 90 and 120 pre-meal, 150, 180, 210, 240 and 300 min post-meal. Metabolic rate was measured every 30 min after each blood sample. Participants were presented to a standard isocaloric PKU type meal at 120 min. After the completion of the last measurement, the participants were presented with an ad libitum buffet test meal.
  Interventions: Other: PKU type meal

INTERVENTIONS:
Other: PKU type meal and Exercise — * Exercise was conducted prior to PKU type meal.
  * PKU type meal was based on PKU special low protein foods (50% of total energy intake), natural free protein foods (37%) and protein substitute (13%). Calories provided in breakfast were 600 kcal and were not based on individual dietary requirement. 65% of total energy intake was provided from carbohydrate, 13% from protein and 22% from fat.
  Arms: Exercise trial
Other: PKU type meal — PKU type meal was based on PKU special low protein foods (50% of total energy intake), natural free protein foods (37%) and protein substitute (13%). Calories provided in breakfast were 600 kcal and were not based on individual dietary requirement. 65% of total energy intake was provided from carbohydrate, 13% from protein and 22% from fat.
  Arms: Control trial

SUMMARY:
The study applied a randomized, crossover design with preliminary (screening) session and two sequenced experimental trials. Trials were marked as Control trial and Exercise trial. Participants were asked to either resting (Control trial) or exercising (Exercise trial) for one hour. In the two trials, appetite questionnaires were obtained, blood samples were collected, and metabolic rates were measured every 30 minutes. Participants in both trials were presented to a standard isocaloric PKU type meal at 120 min. After the completion of the last measurement, the participants were presented with an ad libitum buffet test meal at 300 min. Participants required to record their EI for the remainder of the experimental day using a self-recorded food diary. Two days prior the experimental trials participants refrained from exercise and alcohol intake. All data collection took place in the metabolic research unit at New Lister Building, Glasgow Royal Infirmary.

DETAILED DESCRIPTION:
Participants of the study were essentially healthy men with body mass index (BMI) ≤29 kg/m2 and aged between 22-35 years, recruited by advertisements and word of mouth. Study participants were required to be non-smokers, to have stable body weight for one month prior to study enrolment, and were not taking any medication, nutritional supplement or being on a special diet. Exclusion criteria included chronic illness, eating disorder and history of gastrointestinal operations which could interfere with the results of the study. Written informed consent were obtained prior commencing the study. The Ethics Committee of the collage of Medical Veterinary and Life Sciences, Glasgow University approved the study.

Preliminary session

Before joining the study, preliminary session was conducted for ~3 hours. Participants were informed to come to the metabolic research unit at New Lister Building, Glasgow Royal Infirmary to completed physical activity readiness questionnaire (PARQ), healthy screening questionnaire and International physical activity questionnaire. Only participants at light or moderate of physical activity level, answered "no" to all questions in PARQ and were in generally good health were eligible to complete the preliminary session. Subsequently, height and body mass were measured and a ~30 min submaximal exercise test was conducted at gradually increasing inclines. After 4 minutes of warming up period (3.5 km/hr and 0% incline), participants were walking at a constant speed of 6 km/hr with incline being increased by 2% every 4 min. The test was terminated when the heart rate (HR) reached 85% of maximal HR (HRmax) defined as 220 - age in years. During the test, participants were wearing a HR monitor and a face mask (to measure rate of oxygen consumption (V̇O2) and rate of carbon dioxide production (V̇CO2)). The HR monitor and the mask were both connected to the indirect calorimetry machine (Quark RMR®, COSMED, Italy). The obtained data was used to predict maximal oxygen consumption (V̇O2max) which was achieved by extrapolation of the HR against V̇O2 in order to calculate workload corresponds to 60% of V̇O2max.

Experimental trials

A randomisation scheme was generated using GraphPad Software 2018© to allocate participants to the experimental trials. Trials were marked as Control and Exercise by the researcher. Each participant started first trial according to allocated trial randomization. On the morning of each experiment trial, participants reported to the metabolic research unit between 08:00 and 09:00 after an overnight fast. Height, body mass and resting metabolic rate (RMR) were measured. A cannula was introduced into an antecubital vein and after an interval of 10 min, a baseline blood sample was obtained. Subsequently, an appetite questionnaire was completed. Participants were then asked to either resting (Control trial) or exercising (Exercise trial) for one hour. The Exercise trials were conducted under controlled laboratory conditions. Participants were exercising on the treadmill (Trackmaster Treadmills, Full Vision, Inc., Kansas, USA) at speed and grade corresponding to 60% of their V̇O2max. Participants were wearing a HR monitor and a face mask while exercising, connected to indirect calorimetry equipment (Quark RMR®, COSMED, Italy). V̇O2 and V̇CO2 in the inspired and expired air were measured to calculate fat and CHO oxidation and rate of physical activity energy expenditure (PAEE) by using indirect calorimetry equations described by Frayn and Macdonald (1997).

Subsequently, participants in both trials were presented to a standard isocaloric PKU type meal at 120 min. PKU meals in Exercise and Control trials were matched for weight content and macronutrient composition. Participants were asked to consume the entire meal within 20 min. Appetite questionnaires were obtained and blood samples were collected at 30, 60, 90 and 120 pre-meal, 150, 180, 210, 240 and 300 min post-meal. Metabolic rate was measured every 30 min after each blood sample. After the completion of the last measurement, the participants were presented with an ad libitum buffet test meal which used to assess, under laboratory conditions, the spontaneous macronutrient and energy intake (EI). After completion of each trial, participants required to record their EI for the remainder of the experimental day using a self-recorded food diary. Water was available throughout the trials, but intake was replicated in the second trial and consumption time was matched. During the two days before the first trial, participants weighed and recorded all foods and drinks consumed and were asked to replicate this intake during the two days preceding the second trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men with
* Body mass index (BMI) ≤29 kg/m2
* Aged 22-35 years
* Stable body weight for one month prior to study enrolment, and were
* Not taking any medication, nutritional supplement or being on a special diet.

Exclusion Criteria:

* Smokers
* Chronic illness
* Eating disorder
* History of gastrointestinal operations which could interfere with the results of the study

Ages: 22 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We decided to study males since in case of females the wash out period of approximately 1 month will be needed to ensure that experimental trials are conducted during the same phase of the menstrual cycle.
Enrollment: 16 (Actual)
Dates: Start 2018-06-03 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-07-05 (Actual)

PRIMARY OUTCOMES:
Peptide YY (PYY) | 300 minutes through study completion, an average of 12 days
  Changes in plasma concentration of fasting and postprandial PYY were measured during the Exercise and Control trials.
Glucagon-like peptide-1 (GLP-1) | 300 minutes through study completion, an average of 12 days
  Changes in plasma concentration of fasting and postprandial GLP-1 were measured during the Exercise and Control trials.

SECONDARY OUTCOMES:
Subjective appetite score | 300 minutes through study completion, an average of 12 days
  Appetite scores during Exercise and Control trials were assessed using a 100-mm Visual Analog Scale, with 0 mm meaning one and 100 mm another extreme of hunger, desire to eat, fullness, prospective food consumption, and satiety.
Dietary intake | 24 hours through study completion, an average of 12 days
  Energy and macronutrient intake during Exercise and Control trials was analysed using WinDiets software based on food composition tables.
Diet induced thermogenesis | 300 minutes through study completion, an average of 12 days
  Metabolic rate measured during Exercise and Control trials by means of indirect calorimetry
Growth differentiation factor 15 (GDF-15) | 300 minutes through study completion, an average of 12 days
  Changes in plasma concentration of fasting and postprandial GDF-15 were measured during the Exercise and Control trials.
Fat oxidation | 300 minutes through study completion, an average of 12 days
  Rate of fat oxidation during Exercise and Control trials was measured by means of indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Malkova, PhD, Study Chair — University of Glasgow
Locations (1):
- Univesrity of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No